CLINICAL TRIAL: NCT07247084
Title: A Phase 4 Multicenter, Randomized, Open-Label, Interventional Study With Pragmatic Elements Investigating the Effectiveness of Tirzepatide Once Weekly Compared With Standard of Care in Adult Participants With Obesity and Without Diabetes in a Real-World Setting
Brief Title: A Study of Tirzepatide (LY3298176) Compared With Standard of Care in Adult Participants With Obesity and Without Diabetes (SURMOUNT-REAL UK)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27331; I8F-MC-GPJF (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obesity
Keywords: Overweight; Electronic health records; Primary care; Type 2 diabetes incidence; Obesity related complications; Pragmatic trial; Randomized trial
MeSH Terms: conditions — Obesity; Overweight | interventions — Tirzepatide; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide + Standard of Care (Experimental): Participants will receive tirzepatide subcutaneously (SC) + standard of care
  Interventions: Drug: Tirzepatide
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: Tirzepatide + Standard of Care
Other: Standard of Care — Standard of care
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to evaluate tirzepatide within a real-world setting to assess body weight loss and incidence of type 2 diabetes in adults without diabetes who have obesity and at least one weight-related comorbid condition. Participation in the study will last about 260 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index ≥30 and ≤34.9 kilogram per square meter (kg/m2)
* Have an increased waist to height ratio (defined by >0.5)
* Have at least one weight related comorbid condition
* Have had at least one attempt to lose weight with lifestyle intervention (diet and physical activity)

Exclusion Criteria:

* Have type 1 diabetes, type 2 diabetes, or any other types of diabetes
* Have had a change in body weight of greater than 5 kilograms (11 pounds) within 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, 24 months

SECONDARY OUTCOMES:
Time from Baseline to Onset of Type 2 Diabetes | Baseline through 60 months
Percentage of Participants Converting from Prediabetes to Normoglycemia | 60 months
Percentage of Participants with Normoglycemia at Baseline who Develop Prediabetes | 60 months
Change from Baseline in Hemoglobin A1c (HbA1c) | Baseline, 60 months
Percentage of Participants who Develop a New Obesity-Related Complication | 60 months
Change from Baseline in Waist Circumference | Baseline, 60 months
Change from Baseline in Waist-to-Height Ratio | Baseline, 60 months
Change from Baseline in Total Cholesterol | Baseline, 60 months
Change from Baseline in Systolic Blood Pressure | Baseline, 60 months
Change from Baseline in Diastolic Blood Pressure | Baseline, 60 months
Percent Change from Baseline Urinary Albumin-to-Creatinine Ratio (UACR) | Baseline, 60 months
Change from Baseline in EQ-5D-5L | Baseline, 60 months
Change from Baseline in Impact of Weight on Quality of Life-Lite-Clinical Trials (IWQOL-lite-CT) | Baseline, 60 months
Change from Baseline in Healthcare Resource Utilization (HCRU) | Baseline, 60 months
Change from Baseline in Alanine Aminotransferase (ALT) | Baseline, 60 months
Change from Baseline in Aspartate Aminotransferase (AST) | Baseline, 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (24):
- United Kingdom (24):
  - P91604 St John's Medical Centre, Altrincham
  - P89008 Ashton Medical Group, Ashton-under-Lyne
  - Y02319 SSP Bolton General Practice, Bolton
  - P83012 Tower Family Healthcare, Bury
  - P91014 Washway Road Medical Centre, Cheshire
  - P88007 Cheadle Hulme Medical Group (was Cheadle Hulme Health Centre) (Bridge House), Cheshire
  - Y02790 SSP Bolton Medical Centre, Great Lever
  - P89002 The Brooke Surgery, Hyde SK14
  - P84035 Bodey Medical Centre, Manchester
  - P84630 The Arch Medical Practice, Manchester
  - P86004 Peterloo Medical Centre, Manchester
  - P87019 Silverdale Medical Practice, Manchester
  - P91006 Urmston Group Practice, Manchester
  - P84046 Cheetham Hill Medical Centre, Manchester
  - P92620 SSP Ince Surgery (Lower Ince), Manchester
  - P85010 Woodlands Medical Practice, Oldham
  - P85011 CH Medical Practice, Oldham
  - P86022 Stonefield Street Surgery, Rochdale
  - P91021 Firsway Health Centre, Sale
  - P87027 Langworthy Medical Practice, Salford
  - P88632 Stockport Medical Group, Stockport
  - P87016 The Sides Medical Centre, Swinton
  - P87025 The Lakes Medical Practice, Swinton
  - Y02322 SSP Leigh Family Practice, Wigen

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/